CLINICAL TRIAL: NCT04236674
Title: Thermomechanical Distraction and Social Anesthesia in Interventional Radiology to Improve Patient Satisfaction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TempleU25969
Record Dates: First submitted 2020-01-16; First posted 2020-01-22 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Pain; Analgesia; Anxiety
Keywords: Distraction; Thermomechanical analgesia; Music; Anxiety; Pain; Analgesia; Buzzy; Interventional radiology; IR; Picc; Paracentesis
MeSH Terms: conditions — Pain; Agnosia; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- No intervention (No Intervention)
- Buzzy (Experimental): Thermomechanical device for periprocedural analgesia
  Interventions: Device: Buzzy thermomechanical device
- Music Selection (Experimental): Patient specified music selection for procedural room
  Interventions: Behavioral: Music Selection
- Buzzy and Music Selection (Experimental): A combination of use of the Buzzy device and patient specified music selection
  Interventions: Device: Buzzy thermomechanical device; Behavioral: Music Selection

INTERVENTIONS:
Device: Buzzy thermomechanical device — Buzzy thermomechanical device placed near intervention site.
  Arms: Buzzy; Buzzy and Music Selection
Behavioral: Music Selection — Patient specified procedural music
  Arms: Buzzy and Music Selection; Music Selection

SUMMARY:
The study will prospectively analyze the analgesic and anxiolytic effects of thermomechanical stimulation (cold and vibration effects) with or without patient selected music preference during non-sedating interventional radiology procedures.

DETAILED DESCRIPTION:
There are wide ranging influences on the perception of human pain. The perception of pain is shaped by physiology, genetic factors, prior experiences, and external ameliorating factors. Extensive research has been performed in the pediatric population utilizing distraction as a means of reducing pain, particularly during venipuncture. These methods include medications (i.e. creams, anxiolytics), behavioral distraction (i.e. music, games), cold anesthesia, and thermomechanical stimulation via a cooling/vibrating device; however, fear and anxiety associated with needle procedures does not always resolve with time or age and can result in avoidance of treatment and delays in care. Few studies have focused on the impact of non-pharmacologic anxiolytics using thermomechanical stimulation and social anesthesia (i.e. music as a form of distraction) in the adult population. Utilizing non-pharmacologic measures is one of the first steps in procedural pain management. A thermomechanical device used in the pediatric population called Buzzy (MMJ Labs, Atlanta GA) employs a battery operated, handheld plastic device with a vibrating motor and a mechanism to attach an ice pack. This is used either independently or in combination. Most reports of the device demonstrate significant pain relief, but the majority of these completed studies focused on children undergoing venous cannulation. There have been a few cited uses in adult podiatry, dermatology, and pain management. In addition, passive music based intervention have been used in cancer patients undergoing biopsy and surgery, revealing a significant pain reduction effect. The study will prospectively analyze the analgesic and anxiolytic effects of thermomechanical stimulation (cold and vibration effects) with or without patient selected music preference during non-sedating interventional radiology procedures.

ELIGIBILITY:
Inclusion Criteria:

* 18-90 years of age

Exclusion Criteria:

* prisoners, elderly, minors, pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2020-01-27 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Pain visual analog scale - pre-procedure | Baseline (Prior to the procedure)
  VAS pre-procedure , patient reported, rated 0-100mm with 100mm as the most pain imaginable
Anxiety visual analog scale - pre-procedure | Baseline (Prior to the procedure)
  VAS pre-procedure, patient reported, rated 0-100mm with 100mm as the Worst anxiety
Pain visual analog scale - post-procedure | Immediately after the procedure
  VAS post-procedure , patient reported, rated 0-100mm with 100mm as the most pain imaginable
Anxiety visual analog scale - post-procedure | Immediately after the procedure
  VAS post-procedure, patient reported, rated 0-100mm with 100mm as the Worst anxiety

SECONDARY OUTCOMES:
Satisfaction survey | Immediately after the procedure
  Patient reported satisfaction survey post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ryan M Cobb, MD, Study Director — Temple University Hospital
Locations (1):
- Ryan Michael Cobb, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No